CLINICAL TRIAL: NCT00625417
Title: Breast Tumor Detection Using Optical Spectroscopy
Brief Title: Optical Spectroscopy in Evaluating Tumor Margins in Patients Who Have Undergone Surgery for Breast Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anita Mahadevan-Jansen, Professor, Biomedical Engineering, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000587230; P30CA068485 (NIH); VU-VICC-BRE-0718 (Other Grant/Funding Number: VICC); VU-VICC-060554 (Other Grant/Funding Number: VICC)
Record Dates: First submitted 2008-02-27; First posted 2008-02-28 (Estimated); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
Keywords: male breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male

STUDY DESIGN:
Intervention Model Description: Optical spectroscopy is applied to evaluate tumor margins in consenting patients who undergo surgery for breast tumors

ARMS (1):
- Optical spectroscopy on tumor margins (Experimental): Optical spectroscopy is performed on breast tumor margins obtained from patients undergoing surgery
  Interventions: Procedure: breast biopsy; Procedure: histopathologic examination; Procedure: light-scattering spectroscopy; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Procedure: breast biopsy
Procedure: histopathologic examination
Procedure: light-scattering spectroscopy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Diagnostic procedures, such as optical spectroscopy, may help learn the extent of disease and allow doctors to plan better treatment.

PURPOSE: This phase I trial is studying optical spectroscopy to see how well it works in evaluating tumor margins in patients who have undergone surgery for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To develop a non-invasive detection tool that evaluates breast tumor margins in real-time to guide tumor resection during partial mastectomy procedures.
* To conduct an ex vivo optical spectroscopic study in operating rooms on breast tissue samples obtained immediately following resection to assess the efficacy of using this tool in differentiating breast tumor or tumor margins from normal breast tissue.

OUTLINE: Breast tissue samples obtained immediately following resection are examined in the operating room using optical spectroscopy to evaluate the margin tissue. During spectroscopy, all lights, except for the surgical lights, are turned off and the lateral, superior, medial, inferior, deep, and anterior margins of the breast tissue sample are examined using a fiber-optic probe, a nitrogen laser, and a broad band white light source. Reflectance and fluorescence spectra are measured at each of these margins by a system operator. The measured margins are then immediately marked by sutures placed by the surgeon. Additional margins may be measured at the surgeon's and system operator's discretion. The breast tissue sample is then delivered to surgical pathology, where shave biopsies are performed at the suture-marked sites to provide a direct correlation between spectroscopy measurements and tissue pathology.

Data collected in this study, including spectral data, gross diagnosis of the patient's tumor, and histological identities of all specimens collected, will be kept in the research record for at least 6 years after the study is finished.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Scheduled to undergo lumpectomy, partial or radical mastectomy, or excisional biopsy for breast tumor at Vanderbilt University Hospital
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* Not pregnant

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

INCLUSION CRITERIA Only adult patients between the ages of 18-99 years with breast tumor undergoing lumpectomy, radical mastectomy or excisional biopsy procedure will be considered

EXCLUSION CRITERIA Pregnant women will be excluded from the participation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Development of a non-invasive detection tool that evaluates breast tumor margins in real-time to guide tumor resection during partial mastectomy procedures | 1 year
  A 3-D scanner that can scan a breast lump will be developed so that breast margin may be evaluated with Raman spectroscopy
Evaluated optical spectroscopy in differentiating breast tumor or tumor margins from normal breast tissue | 2 years
  This device will be tested in patient specimens intra-operatively before going to pathology and compared to histopathology to evaluate the ability of the device to detect margin up to 2 mm deep

CONTACTS AND LOCATIONS:
Overall Officials: Anita Mahadevan-Jansen, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
This is still an early phase study and the data is not ready for dissemination yet.